CLINICAL TRIAL: NCT02803736
Title: Effectiveness of Acupuncture for Breast Cancer Related Lymphedema
Acronym: Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fourth Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Liuzhou Hospital of Traditional Chinese Medicine (Other); Liuzhou Maternity and Child Healthcare Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJK201690
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer; Lymphedema; Acupuncture
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real acupuncture group (Experimental): Patients in the real acupuncture group will receive true acupuncture 3 times a week for 4 weeks (12 sessions). A standardized prescription of six acupuncture points is used unilaterally. Needles are inserted and manipulated manually until needling sensation (de qi) is obtained, and are retained for 20 minutes with manual manipulation at 10 minutes. Acupuncturists are trained to inquire about specific needle sensations when providing true acupuncture.
  Interventions: Device: acupuncture
- Sham acupuncture group (Sham Comparator): Patients in the sham acupuncture group will receive sham acupuncture 3 times a week for 4 weeks (12 sessions).
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — Acupuncture involves the insertion of extremely thin needles through skin at strategic points on human body. Many Western practitioners view the acupuncture as a device to stimulate nerves, muscles and connective tissue, and believe that it can increases blood flow.
  Other Names: zhen jiu

SUMMARY:
This multicenter placebo-controlled trial focuses on the efficacy and safety of acupuncture on breast-cancer related lymphedema. 200 participants will be recruited, and randomized in two groups: the real acupuncture group and the sham acupuncture group.

DETAILED DESCRIPTION:
In the theory of Traditional Chinese Medicine (TCM), Breast Cancer Related Lymphedema (BCRL) is classified as "edema", and is considered to be caused by qi (chi) deficiency and blood stagnation. Acupuncture, as an ancient therapy in TCM, is thought to have the efficacy to stimulate the transformation of qi and drainage of dampness, and is widely used for various diseases including edema in China. Early clinical trials as well as our own clinical observation have demonstrated that acupuncture can ameliorate limb swelling and decrease lymphedema. However, no randomized placebo-controlled trial has been performed to evaluate this efficacy of acupuncture. Therefore, this study aimed to evaluate the safety and potential efficacy of acupuncture to treat chronic upper-limb lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* women who completed all primary and adjuvant treatments.
* age between 20 and 45.
* BMI between 18 and 28.
* unilateral lymphedema resulting from surgery for breast cancer.
* mild to moderate lymphedema, with 10% to 40% increase in volume compared to the unaffected arm based on perometry evaluation.
* with no evidence of recurrence.

Exclusion Criteria:

* bilateral lymphedema.
* history of bilateral axillary lymph node dissection.
* serious lymphedema, with over 40% increase in volume compared to the unaffected arm based on perometry evaluation.
* pregnant women.
* unable to adhere to the protocol or the treatment schedule.
* recurrent breast cancer or other malignancies.
* current use of chemotherapy or radiation.
* current use of diuretic drugs like Diosmin, or other investigational drugs.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Absolute Reduced Limb Volume Ratio | Day 0 (baseline), Day 30(endpoint)
  Data of the absolute limb volume will be collected before the treatment (volume at baseline, B) and after the treatment (volume after therapy, A) for every participant. VL is the volume of the affected arm with lymphedema, and VC is the volume of the contralateral arm. Then, The ARLVR will be calculated using the following formula: ARLVR (%) = (VL-Vc)B-( VL-Vc)A/( VL-Vc)B ×100%.
  The arm measurement will be conducted using perometer. This method is inspired by the method established by Anderson et al.

SECONDARY OUTCOMES:
Incidence of Adverse Event | Day 0 (baseline), Day 30(endpoint)
  Every adverse event during the treatment will be recorded, unless it is confirmed otherwise, whereas those occurs after the treatment will not be calculate unless it is confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Wei, Principal Investigator — Guangxi Medical University Institutional Review Board

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersen L, Hojris I, Erlandsen M, Andersen J. Treatment of breast-cancer-related lymphedema with or without manual lymphatic drainage--a randomized study. Acta Oncol. 2000;39(3):399-405. doi: 10.1080/028418600750013186. PMID 10987238
- [Derived] Zhu H, Li J, Peng Z, Huang Y, Lv X, Song L, Zhou G, Lin S, Chen J, He B, Qin F, Liu X, Dai M, Zou Y, Dai S. Effectiveness of acupuncture for breast cancer related lymphedema: protocol for a single-blind, sham-controlled, randomized, multicenter trial. BMC Complement Altern Med. 2017 Sep 21;17(1):467. doi: 10.1186/s12906-017-1980-0. PMID 28934950